CLINICAL TRIAL: NCT00053118
Title: High Dose Carboplatin Combined With Oral VP-16 In The Treatment Of Pediatric CNS Malignancies
Brief Title: Chemotherapy and Stem Cell Transplantation in Treating Children With Central Nervous System Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Barbara Bambach, MD, Roswell Park Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000269284; RPCI-DS-00-03
Record Dates: First submitted 2003-01-27; First posted 2003-01-28 (Estimated); Last update posted 2011-03-01 (Estimated); Status verified 2011-02

CONDITIONS: Brain and Central Nervous System Tumors; Lymphoma; Neuroblastoma; Retinoblastoma
Keywords: childhood central nervous system germ cell tumor; childhood choroid plexus tumor; childhood craniopharyngioma; childhood grade I meningioma; childhood grade II meningioma; childhood grade III meningioma; recurrent childhood brain stem glioma; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma; recurrent childhood ependymoma; recurrent childhood medulloblastoma; recurrent childhood supratentorial primitive neuroectodermal tumor; recurrent neuroblastoma; recurrent retinoblastoma; childhood visual pathway and hypothalamic glioma; childhood atypical teratoid/rhabdoid tumor; primary central nervous system non-Hodgkin lymphoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Lymphoma; Neuroblastoma; Retinoblastoma; Choroid Plexus Neoplasms; Astrocytoma; Familial ependymoma; Medulloblastoma; Optic Nerve Glioma; Rhabdoid Tumor | interventions — Filgrastim; Carboplatin; Etoposide; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: filgrastim — IV
Drug: carboplatin — IV
Drug: etoposide — IV
Procedure: bone marrow ablation with stem cell support — IV
Procedure: peripheral blood stem cell transplantation — IV

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining chemotherapy with peripheral stem cell transplantation in treating children who have central nervous system cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of administering an outpatient protocol comprising high-dose carboplatin with autologous stem cell support and etoposide in pediatric patients with primary central nervous system malignancies.
* Determine the maximum tolerated dose of carboplatin when administered in this regimen in these patients.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is dose-escalation study of carboplatin.

Patients receive filgrastim (G-CSF) IV once daily for 6 days followed by a maximum of 5 apheresis sessions. If the target number of peripheral blood stem cells is not achieved, some patients receive G-CSF and undergo apheresis as above after a 2-week rest.

At least 3 days after completion of G-CSF, patients receive high-dose carboplatin IV over 1 hour on day 1, stem cell reinfusion on day 3, G-CSF subcutaneously on days 4-18 and 43-61, and oral etoposide 3 times daily on days 21-42. Treatment continues for a maximum of 4 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of carboplatin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed monthly for 1 year and then annually thereafter.

PROJECTED ACCRUAL: A total of 3-15 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary central nervous system malignancy
* Recurrent, persistent, or progressive disease after at least 1 prior first-line treatment regimen

PATIENT CHARACTERISTICS:

Age

* 18 and under at initial diagnosis

Performance status

* ECOG 0-2

Life expectancy

* At least 8 weeks

Hematopoietic

* Absolute neutrophil count greater than 750/mm^3
* WBC greater than 2,500/mm^3
* Platelet count greater than 100,000/mm^3
* No underlying myelodysplasia, stem cell disorder, or other inherent hematologic synthetic defect

Hepatic

* Liver function tests less than 2 times normal OR
* Absence of active hepatitis by liver biopsy
* Bilirubin less than 1.5 mg/dL

Renal

* Glomerular filtration rate greater than 60 mL/min by radionucleotide assay

Cardiovascular

* Ejection fraction at least 45%

Pulmonary

* Clinically normal pulmonary function (patients 5 years of age and under)
* FEV_1 and FVC at least 50% (patients over 5 years of age) OR
* Arterial blood gas normal and DLCO greater than 50%

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No mucositis or mucosal infection
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* At least 3 weeks since prior systemic cytotoxic chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* At least 6 months since prior radiotherapy to the pelvis or spine

Surgery

* Not specified

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2002-03; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Jean Bambach, MD, Study Chair — Roswell Park Cancer Institute
Locations (3):
- United States (3):
  - St. Louis Children's Hospital, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of Texas - MD Anderson Cancer Center, Houston, Texas